CLINICAL TRIAL: NCT01505790
Title: Impact of Clopidogrel Dose Adjustment According to Platelet Reactivity Monitoring in Patients With High on Treatment Platelet Reactivity Undergoing Percutaneous Coronary Intervention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-020095-32; 2009-39 (Other: AP HM)
Record Dates: First submitted 2011-08-25; First posted 2012-01-09 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Acute Coronary Syndromes
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CLOPIDOGREL GROUP (Experimental)
  Interventions: Drug: Clopidogrel
- PRASUGREL GROUP (Active Comparator)
  Interventions: Drug: PRASUGREL

INTERVENTIONS:
Drug: PRASUGREL — 60 mg the first day then 10 mg per day during one month
  Arms: PRASUGREL GROUP
Drug: Clopidogrel — 600 mg clopidogrel will be administered during the first 6 to 12 hours then a measure of platelets reactivity will be done. An additional administration of clopidogrel (600 mg) could be done every 6 hours until to obtain a VASP <50%. No more than 3 * 600mg of clopidogrel will be authorized in this protocol.
  Then for patient which have received more than one dose of clopidogrel 600mg , 150 mg per day of clopidogrel will be administrated, for which who have received only one dose of 600mg of clopidogrel , 75 mg per day will be administrated during one month at least.
  Arms: CLOPIDOGREL GROUP

SUMMARY:
Acute coronary syndromes are related to the development of a platelet derived thrombus on a ruptured coronary atheroma. Use of dual antiplatelet therapy aspirin-thienopyridine a significantly reduced the risk of major adverse cardiovascular events (MACE) after percutaneous coronary intervention (PCI). However despite these therapeutic innovations, the rate of MACE in patients treated using PCI and particularly in those suffering of an acute coronary syndrome is around 5% in randomized trials. Within the factors associated with MACE, high on treatment platelet reactivity following clopidogrel loading dose has been identified as a key factor. In fact it is widely recognized that there is a large inter individual variability in clopidogrel responsiveness. In addition several authors have demonstrated a strong link between high on treatment platelet reactivity following clopidogrel loading dose and the occurrence of post PCI MACE. Vasodilator Phosphoprotein index measurement (VASP index) enables a reproducible, standardized and specific assessment of clopidogrel responsiveness.

The investigators previous works have demonstrated that a VASP index ≥ 50% had a high negative predictive value for post PCI MACE in patients undergoing PCI and that tailored clopidogrel loading dose in order to obtain a VASP index < 50% before PCI resulted in a reduction in the rate of post PCI MACE.

Prasugrel is a new generation thienopyridine with a faster and more powerful anti platelet effect compared to clopidogrel. It was shown to be superior to clopidogrel to reduce post PCI MACE in acute coronary syndromes. However in this randomized trial prasugrel achieved an excessive blockade of platelet reactivity responsible for a significant increase in bleeding events in some patients and an insufficient blockade in up to 325% of the remaining patients.

Therefore the investigators hypothesized that a strategy of individually tailored loading and maintenance dose of clopidogrel may be superior to prasugrel standard therapy in achieving an optimal platelet reactivity inhibition in acute coronary syndrome patients undergoing PCI.

ELIGIBILITY:
Inclusion Criteria:

* Subject in front of benefited from a coronary angioplasty with setting-up of an endoprothese for a SCA
* Subject agreeing to be followed over a period of 1 month
* Subject agreeing to participate in the research and having given its signed enlightened consent

Exclusion Criteria:

* Subject minor or of more than 75 years old

  * Subject presenting a rate of red blood cells < 4 G/l or a thrombocytopenia > 100 000 / mm3 plaques
  * unaffiliated Subject in a benefit system
  * pregnant or breast-feeding Woman: a pregnancy test will be realized in a systematic way, as well as a stake under contraception of the women old enough to procreate
  * Intolerance or allergy in the aspirin or in the clopidogrel
  * Pathology associated with a life expectancy 6-month-old subordinate according to the investigator
  * haemorrhagic Syndrome threatening the vital forecast, the intra-cranial tumor
  * Contraindication in one of the medicines of the study
  * Severe hepatocellular incapacity
  * Fibrinolyse meadow or hospital intra
  * Ceaseless ventricular arrhythmias
  * State of cardiogenic shock
  * History of cerebral vascular accident
  * Weight lower than 60 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
the biological efficacy of tailored clopidogrel therapy | 12 months
  To compare the biological efficacy of tailored clopidogrel therapy according to the VASP index and prasugrel standard therapy in acute coronary syndromes patients undergoing PCI.

SECONDARY OUTCOMES:
clinical efficacy | 12 MONTHS
  Baseline in Systolic Blood Pressure at 6 months
Tolerability | 12 MONTHS
  adverse event outcome at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France